CLINICAL TRIAL: NCT01085578
Title: Evaluation of Safety,Tolerability and Pharmacokinetic Characteristics of CG400549 in Healthy Volunteers
Brief Title: CG400549 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CG400549-1-01
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: healthy male volunteers; fasted and fed state
MeSH Terms: interventions — CG 400549; KPNA1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort1 (Placebo Comparator): CG400549/placebo
  Interventions: Drug: CG400549/placebo
- Cohort2 (Placebo Comparator): CG400549/placebo
  Interventions: Drug: CG400549/placebo
- Cohort3 (Other): CG400549
  Interventions: Drug: CG400549

INTERVENTIONS:
Drug: CG400549/placebo — Period 1: a single oral dose of 80 mg CG400549 or placebo on Day 1 Period 2: a single oral dose of 320 mg CG400549 or placebo on Day 1 Period 3: a single oral dose of 1280 mg CG400549 or placebo on Day 1
  Other Names: Cohort 1
  Arms: Cohort1
Drug: CG400549/placebo — Period 1: a single oral dose of 160 mg CG400549 or placebo on Day 1 Period 2: a single oral dose of 640 mg CG400549 or placebo on Day 1 Period 3: a single oral dose of 1920 mg CG400549 or placebo on Day 1
  Other Names: Cohort 2
  Arms: Cohort2
Drug: CG400549 — Period 1: a single oral dose of 640 mg CG400549 on Day 1 in the fasted state Period 2: a single oral dose of 640 mg CG400549 on Day 1 in the fed state
  Other Names: Cohort 3
  Arms: Cohort3

SUMMARY:
Evaluation of Safety, Tolerability and Pharmacokinetic Characteristics of CG400549 in Healthy Volunteers

DETAILED DESCRIPTION:
This was a Phase 1, 2-part study consisting of a randomized, double-blind, placebo-controlled,single ascending dose (SAD) part (in 2 alternating panels) and a 1-sequence food effect (FE) part. In the SAD part, 2 cohorts of 6 healthy male subjects each received a single oral dose of CG400549 or placebo in 3 periods, randomized such that each subject received active treatment twice and placebo once (in each period, 4 subjects received active drug and 2 received placebo). In the FE part, 1 cohort of 6 healthy male subjects received a single oral dose of CG400549 in the fasted state in Period 1 and a single oral dose of CG400549 in the fed state in Period 2.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sex : male
* 2. Age : 18-55 years, inclusive
* 3. BMI : 19-30 kg/m2
* 4. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks"), grapefruit (juice) and tobacco products from 48 h prior to entry in the clinical research centre until discharge
* 5. Medical history without major pathology
* 6. Normal blood pressure (systolic 90-140 mmHg; diastolic 60-90 mmHg) and heart rate (45 90 beats per minute); minor deviations from these criteria could be accepted if considered to be clinically insignificant by the Medical Investigator
* 7. Computerised (12-lead) ECG recording normal or showing no clinically relevant deviations as judged by the Medical Investigator
* 8. Male subjects and their female sexual partners must use double-barrier contraception during the study period and for 90 days after follow-up
* 9. All values for haematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Medical Investigator. In particular, liver enzymes (aspartate aminotransferase [ASAT] and alanine aminotransferase [ALAT]) must be within the normal range and creatine phosphokinase (CPK) must be within 2.0 times the normal range.
* 10. Willingness to sign the written Informed Consent Form (ICF)

Exclusion Criteria:

* 1. Evidence of clinically relevant pathology
* 2. History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 1 month of study
* 3. Presence or history of esophageal or gastroduodenal ulceration within 1 month before screening.
* 4. Family history of significant cardiac disease (e.g., sudden cardiac death or myocardial infarction prior to age 50 in a first-degree relative)
* 5. Mental handicap, relevant cognitive or psychiatric disorders or history of seizures
* 6. History and/or presence of relevant drug and/or food allergies
* 7. Use of concomitant medication, except for acetaminophen (paracetamol), which is allowed up to 3 days before entrance into the research facility. All other medication (including over-the-counter medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to the first dose. The use of a limited amount of acetaminophen (≤ 2 g/day) is permitted.
* 8. Participation in a drug study within 60 days prior to drug administration. Participation in more than 3 other drug studies in the 10 months preceding the start of this study.
* 9. Donation of more than 50 mL of blood (whole blood or blood component) within 60 days prior to drug administration.
* 10. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
* 11. Positive screen on drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids), barbiturates, benzodiazepines, tricyclic antidepressants and alcohol
* 12. Intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
* 13. Positive screen on hepatitis B surface antigen (HBsAg)
* 14. Positive screen on anti hepatitis C virus (HCV)
* 15. Positive screen on anti human immunodeficiency virus 1 and 2 (HIV 1/2)
* 16. Illness within 5 days prior to drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | up to 4 weeks

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration of CG400549 (Cmax) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hour post-dose
Area Under the Concentration-Time Curve of CG400549 (AUC) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36 and 48 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Seonggu Ro, PhD, Study Chair — CrystalGenomics, Inc.
Locations (1):
- PRA International clinical center, Zuidlaren, Netherlands